CLINICAL TRIAL: NCT01461317
Title: A Phase II Open-Label Extension Study to Evaluate the Long-Term Safety of Etrolizumab in Patients With Moderate to Severe Ulcerative Colitis
Brief Title: Study to Evaluate the Long-term Safety of Etrolizumab in Participants With Moderate to Severe Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GA27927; 2011-003409-36 (EudraCT Number)
Record Dates: First submitted 2011-10-12; First posted 2011-10-28 (Estimated); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — etrolizumab

ARMS (1):
- Etrolizumab (Experimental): Etrolizumab 100 milligrams (mg) subcutaneous (SC) administration every 4 weeks during the treatment period of up to 240 weeks.
  Interventions: Drug: Etrolizumab

INTERVENTIONS:
Drug: Etrolizumab — Participants will receive etrolizumab at a dose of 100 mg.

SUMMARY:
This study is an open-label extension (OLE) trial to evaluate the safety and tolerability of etrolizumab in participants with moderate to severe ulcerative colitis (UC) who were enrolled in the Phase II Study ABS4986g (NCT01336465) and meet the eligibility criteria for entry in the OLE study.

ELIGIBILITY:
Inclusion Criteria:

* All participants (placebo or active) who were previously enrolled in the Phase II study (ABS4986g) and fulfill any of the following criteria:
* Participants who have not obtained a clinical response in the Phase II study (ABS4986g) by Week 10 (the end of the Phase II treatment phase) may enter this OLE trial at any time after Week 10 and up to and including Week 28
* Participants who have a clinical response in the Phase II study (ABS4986g) at Week 10 but have had a flare of UC between Week 10 and Week 28
* Males and females with reproductive potential must be willing to use a highly effective method of contraception, vaginal ring, intrauterine device, physical barrier, or vasectomized partner) from study start to a minimum of 4 months (approximately 5 half-lives)
* Concomitant immunosuppressive therapy must be tapered within 6 weeks after enrollment in this OLE study
* Participants must have tapered completely off oral corticosteroids within 24 weeks of enrollment to this OLE study

Exclusion Criteria:

* Participants who did not complete through Week 10 of the Phase II study (ABS4986g)
* Pregnancy or lactation
* Any new malignancy within the past 6 months
* Any new (since enrolling in the Phase II study [ABS4986g]), significant, uncontrolled, co- morbidity, such as neurological, cardiac, pulmonary, renal, hepatic, endocrine, or gastrointestinal (GI) disorders
* Any new clinically significant signs or symptoms of infection as judged by the investigator
* Any abnormal laboratory values recorded at the last visit completed in the Phase II study (ABS4986g)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2011-11-29 (Actual); Primary Completion 2016-08-07 (Actual); Study Completion 2016-08-07 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs) | Baseline up to approximately Week 246
Percentage of Participants With Anti-Therapeutic Antibodies (ATAs) to Etrolizumab | Baseline up to approximately Week 246 (assessed at predose (Hour 0) at baseline, Weeks 4, 8, 12, and every 12 weeks thereafter up to Week 252, 12 weeks after last dose [up to approximately Week 246])

SECONDARY OUTCOMES:
Serum Concentrations of Etrolizumab | Predose (Hour 0) at baseline, Weeks 4, 8, 12, and every 12 weeks thereafter up to approximately Week 246; 12 weeks after last dose (up to approximately Week 246)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (40):
- United States (5):
  - University of California, San Diego, La Jolla, California
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Long Island Clin Rsch Asc, LLP, Great Neck, New York
  - Consultants for Clin. Rsrch, Cincinnati, Ohio
- Australia (4):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - St Vincent's Hospital Melbourne; Department of Gastroenterology, Fitzroy, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital; Gastroenterology, Parkville, Victoria
- Belgium (3):
  - Imeldaziekenhuis, Bonheiden
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
- Canada (4):
  - GI Research Institute, Vancouver, British Columbia
  - London Health Sciences Centre; Victoria Hospital, London, Ontario
  - London Health Sciences Centre, London, Ontario
  - Toronto Digest. Disease Asso., Woodbridge, Ontario
- Czechia (4):
  - Poliklinika Iii, Hk; Hepatogatroenterolgy, Hradec Králové
  - Oblastni nemocnice Nachod a.s.; Endoskopicke centrum, Náchod
  - Fakultni nemocnice Ostrava, Ostrava - Poruba
  - Krajska nemocnice Tomase Bati, Zlín
- Germany (5):
  - CAMPUS VIRCHOW-KLINIKUM; Charité Centrum 13; Med. Klinik Abt. Hepatologie u. Gastroenterologie, Berlin
  - Med. Hochschule Hannover; Gastroenterologie, Hanover
  - Universitatsklinikum Schleswig Holstein; Klinik fur Allgemeine Innere Medizin, Kiel
  - Facharzt für Gastroenterologie, Minden
  - Univ klinikum Ulm; Medizin Zentrum Innere Medizin I, Ulm
- Hungary (3):
  - ENDOMEDIX Kft; Gasztroenterológia Budapest, Budapest
  - Pannónia Klinika Magánorvosi, Budapest
  - Petz Aladar County Hosp; 1St Dept. of Internal Med., Győr
- Israel (5):
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Shaare Zedek Medical Ctr; Dept. of Gastroenterology, Jerusalem
  - The Chaim Sheba Medical Center; Multiple Sclerosis Center, Ramat Gan
  - Tel Aviv Sourasky Medical Ctr; Gastroenterology Department, Tel Aviv
- New Zealand (4):
  - Middlemore Hospital, Auckland
  - University of Otago, Christchurch, Christchurch
  - Dunedin Hospital; Otago District Health Board, Dunedin
  - Shakespeare Specialist Group, Takapuna
- Hospital Clinic I Provincial, Barcelona, Spain
- United Kingdom (2):
  - St. Mark's Hospital; Inflammatory Bowel Disease Unit, Harrow
  - Royal Victoria Infirmary, Newcastle upon Tyne